CLINICAL TRIAL: NCT04166279
Title: The Recovery of Reaching Movement in Breast Cancer Survivors: Two Different Rehabilitative Protocols in Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Doctor, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLS-2019a
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Breast Cancer Lymphedema; Pain; Pain, Postoperative; Pain, Chronic; Mastectomy; Lymphedema; Breast Surgery
Keywords: Breast Cancer; Pain Chronic and Postoperative; Lymphedema; Posture; Target - Reaching movement; Breast surgery; Functional impotence; Rehabilitive treatment; Physiotherapy; Scapula tilting
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema; Pain; Pain, Postoperative; Chronic Pain; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single rehabilitative Treatment (Experimental): Patients treated within single rehabilitative protocol
  Interventions: Other: Single rehabilitative treatment
- Group rehabilitative Treatment (Experimental): Patients treated within group rehabilitative protocol
  Interventions: Other: Group rehabilitative treatment

INTERVENTIONS:
Other: Single rehabilitative treatment — The rehabilitation treatment, performed by a physiotherapist trained in oncological rehabilitation, was carried out with a 6-week exercise program for 12 sessions (60 minutes/session, 2/week).). The protocol included a first phase consist in low impact aerobics warming (15-20 minutes), then diaphragmatic breathing and postural exercises for the midline alignment. The awareness of abdominal breathing represents the preliminary phase for a complete psychophysical relaxation of the patient, an important prerequisite for the correct execution of subsequent mobility, stretching and strengthening exercises of spine, scapula and upper limb. Subsequently, isometric strengthening exercises for shoulder stabilizing muscles, first passively and, subsequently, with supervision, were performed. Specific exercises, for passive mobilization and stabilization of the scapula, cervical pumping and stretching of the pectoral muscles, have been performed.
  Arms: Single rehabilitative Treatment
Other: Group rehabilitative treatment — Four-five patients for group. The rehabilitation treatment, performed by a physiotherapist trained in oncological rehabilitation, was carried out with a 6-week exercise program for 12 sessions (60 minutes/session, 2/week). The protocol included at first week mainly breathing techniques, then we introduced exercises gradually more active, according to the improvements of the execution. The exercises had the aim to improve the opening of the scapular chain and to increase the amplitude of the range of motion in order to stimulate better neuromuscular control during the movement of scapular retropulsion, to stretch the pectoral muscles following the rhythm of the breath and the tissues affected by post-surgical scars and fibrotic effects, finally to reinforcing, against gravity, the musculature of the shoulders and back.
  Arms: Group rehabilitative Treatment

SUMMARY:
This study emphasizes the importance of rehabilitation in breast cancer survivors after mastectomy, even during the course of radiotherapy and chemotherapy, both for good efficacy in reducing pain and for functional recovery of the upper limb. Authors designed a randomized-controlled trial to compare two different rehabilitation protocols: the single rehabilitative treatment (ST) and the group treatment (GT). The study is the first attempt to measure the reaching movement after BC surgery with an optoelectronic evaluation system previously standardized in the neurological field during rehabilitation treatment.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer in women in the developed world. Surgery and medical protocols have improved significantly over the last 10 years and this guarantees a better chance of survival and an improvement in quality of life.

Then, the focus on "what happen after defeating BC" has become current: patients' and physicians' awareness of the sequelae of BC surgery has increased, especially in the case of mastectomy or modified radical mastectomy. A large number of these complications, such as lymphedema or post-treatment pain with or without functional impotence, which contribute to limitations in daily life activities, can be treated favourably and, in sometimes, resolved with early rehabilitation protocols. Therefore, it is not only important to start the rehabilitation process early after surgery, but, also, during the sub-acute phase, choose appropriate exercise programs to allow recovery in "quantity" and "quality" of the movement of the operated upper limb (UL). Alterations in muscle activation and reduced shoulder mobility are common in patients with BC. It is necessary to consider that winged scapula incidence in BC surgery is 8% and the prevalence decreased during 6 months after surgery. In particular, patients who developed winged scapula had more shoulder flexion, adduction and abduction limitation. These findings suggest that, after BC surgery, soft tissues restrictions obstruct short-term scapula motion.

Reaching movement is a complex multi-articular movement towards a defined point in space and allows the hand to interact with the environment. Nevertheless, it is not yet investigated during the rehabilitation process. Moreover, the execution of the UL movements, improves if the numerous perturbations of the musculoskeletal system, which occur during the execution of movements, are compensated. Motor synergy's components should modify their action to influence positively the outcome of motor activity, preventing the mistakes of the individual components from influencing the overall activity. An important issue is represented by the redundancy of the degrees of motor freedom. Actions and movements can be performed in different ways because the functional synergies are able to co-vary, without changing the result of the action. However, only three spatial dimensions are needed to specify any position where the hand could be placed. This excess of kinematic degrees of freedom means that there are multiple arm configurations that correspond to any particular position of the hand. Thus, improvements in reaching, after BC mastectomy, can be determined, compared to a different rehabilitation protocol, by comparing the Single rehabilitative Treatment (ST) with Group Treatment (GT). Authors designed a randomized-controlled trial to check if specific scapula exercises, included in the ST, could induce changes in the fluidity of the reaching, called Jerk (primary outcome), decrease shoulder pain and improve the functioning of the operated upper limb (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* total mastectomy carried out 12 months prior to recruitment for rehabilitation with breast prostheses or tissue expanders performed
* age from 18 to 60 years
* body mass index (BMI) < 30
* no cognitive dysfunctions ( Mini Mental State Examination MMSE > 24)

Exclusion Criteria:

* presence of lymphangitis or mastitis
* presence of metastasis
* surgical complications
* neurological deficits
* shoulder joint problems before surgery
* severe-moderate lymphedema and web axillary syndrome
* visual problem not corrected by lenses

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Change [over time] of the normalized jerk (NJ) within biomechanical reaching movement | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The normalized jerk (NJ) was evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), calculated on the wrist-target marker distance, within the reaching task performed on the side underwent surgery. It measures the fluidity of the upper limb movement.

SECONDARY OUTCOMES:
Change [over time] of Visual Analogue Scale (VAS) | T0 baseline - T1 (6 weeks) - T2 (3 months)
  Instrument to assess unidimensional measure of pain intensity. VAS was presented in a coloured scale with a middle point, graduations and numbers. Under the scale there was a straight horizontal line of fixed length, 100 mm. The ends were defined as the limits of the parameter to be measured (pain in the last 24 hours), orientated from the left (worst, no pain) to the right (best, worst pain to be imagined). The score is determined by measuring the distance (cm) on the 10 cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10.
Change [over time] of Disabilities of Arm, Shoulder and Hand Questionnaire (DASH) | T0 baseline - T1 (6 weeks) - T2 (3 months)
  Self-administered region-specific outcome instrument developed as a measure of self-rated upper-limb disability and symptoms, actually used to monitor changes in symptoms and function over time. It consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The items are related to the degree of difficulty in performing various functional activities because of arm, shoulder or hand limitations (21 items), the intensity of pain, activityrelated pain, tingling, weakness and stiffness (5 items), and the effect related to social activities, job, sleep and its psychological impact (4 items).
Change [over time] of Movement Duration (MD) of biomechanical reaching movement | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The movement duration (MD) was evaluated in seconds, through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery.
Change [over time] of the angle of arm flexion at end of movement (AAF) within biomechanical reaching movement | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The degrees of the angle of arm flexion at end of movement (AAF) were evaluated through the Smart D500 stereophotogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery. A zero value is conventionally assigned to AAF when the arm is along the side, positive values represent flexion, negative ones represent extension.
Change [over time] of the angle at elbow at end of movement (AE) within biomechanical reaching movement | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The degrees of the angle at elbow at end of movement (AE) were evaluated through the Smart D500 stereophotogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery. The value assigned is zero when the elbow is completely extended, positive values correspond to flexion, and negative ones to hyperextension.
Change [over time] of the mean value of target-approaching velocity (TAV) within biomechanical reaching movement | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The mean value of target-approaching velocity (TAV) was evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery.

OTHER OUTCOMES:
Change [over time] of range of Motion (ROM) of shoulder | T0 baseline - T1 (6 weeks) - T2 (3 months)
  The degrees of flexion, extension, adduction, abduction and internal and external rotation evaluated on the side underwent surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Umberto I Hospital, Rome, Italy